CLINICAL TRIAL: NCT06945094
Title: A Multi-center, Real-World Clinical Trial on Assessment of Microcirculatory Status Using Online Coronary Angiography-Derived Index of Microcirculatory Resistance (caIMR) (Flash V)
Brief Title: A Multi-center, Real-World Clinical Trial of caIMR on Two Specific Kinds of Patients.
Acronym: FlashV
Status: Not yet recruiting | Type: Observational
Sponsor: Ge Junbo (Other)
Collaborators: RainMed Medical Group (Industry)
Responsible Party: Sponsor-Investigator, Ge Junbo, Coordinating Investigator, Fudan University
Organization: Fudan University (Other)
Other Study IDs: FlashV
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Coronary Microvascular Dysfunction (CMD); Stable Angina Pectoris; Unstable Angina Pectoris; Myocardial Ischemia, Angina Pectoris
Keywords: Hemodynamics; Computational fluid dynamics; Angiography-derived IMR; coronary microvascular dysfunction; stable and unstable angina
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Myocardial Ischemia; Angina Pectoris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grey zone patients: Patients with caIMR values between 20 and 30 can be enrolled in this group, a total of 254 patients of this type will be enrolled in the study.The binary classification performance of caIMR will be validated based on differences in their Seattle Angina Questionnaire (SAQ) scores and their health outcomes.
  Interventions: Device: caIMR
- Diffuse disease patients.: Patients with diffuse coronary disease and less than 50% stenosis can be enrolled in this group, a total of 254 patients of this type will be enrolled in the study. CaIMR will be assessed in these patients, and its binary classification performance will be validated based on differences in their Seattle Angina Questionnaire (SAQ) scores and their health outcomes.
  Interventions: Device: caIMR

INTERVENTIONS:
Device: caIMR — caIMR will be measured by pressure sensors which are produced by Suzhou Rainmed Medical Technology Co., Ltd.
  caIMR is calculated based on angiography images and Hyperemic Pa estimated from resting Pa according to prespecified equation

SUMMARY:
The coronary angiography-derived index of microcirculatory resistance (caIMR) can be used to provide a binary assessment whether patients（with stable angina, unstable angina, suspected myocardial ischemia, or coronary artery stenosis of less than 50%, and without cardiomyopathy or obstructive epicardial coronary artery disease） have microcirculatory dysfunction, using a cutoff value of 25.

This study aims to evaluate the binary classification performance of caIMR in two specific groups of patients: (1) those with caIMR values between 20 and 30, and (2) those with diffuse disease. We will do this by looking at differences in their Seattle Angina Questionnaire (SAQ) scores and their health outcomes over a three-year period.

DETAILED DESCRIPTION:
The coronary angiography-derived index of microcirculatory resistance (caIMR) is a novel, non-invasive, imaging-based functional index for diagnosing coronary microvascular disease, which has been clinically validated for market release. It can be used to provide a binary assessment of whether patients with stable angina, unstable angina, suspected myocardial ischemia, or coronary artery stenosis of less than 50% (without cardiomyopathy or obstructive epicardial coronary artery disease) have microcirculatory dysfunction, using a cutoff value of 25.

This trial is a prospective, multicenter, observational real-world study. We will regularly collect clinical diagnostic data (including angiographic images) patients who undergo caIMR measurement using the Coronary Artery Functional Measurement System and single-use pressure sensors as part of their routine medical care. After verifying the inclusion and exclusion criteria, patients who meet the inclusion criteria and do not meet the exclusion criteria will be enrolled in this trial.

The primary objective of this trial is to evaluate the binary classification performance of caIMR by comparing patients' Seattle Angina Questionnaire (SAQ) scores before the procedure and at six months post-procedure in two specific groups of patients: :

1. Assessing the binary classification performance of caIMR in patients with values between 20 and 30.
2. Assessing the binary classification performance of caIMR in patients with diffuse disease.

The secondary objective is to validate the prognostic value of caIMR in these two groups of patients based on the occurrence of major adverse cardiovascular events (MACE) over a three-year period.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years, regardless of gender;
2. Diagnosed with stable angina, unstable angina, or suspected myocardial ischemia;
3. targeted vessel stenosis < 50% and caIMR values between 20 and 30; or

(3) Targeted vessel stenosis < 50%, but with lesion length > 20 mm and caFFR > 0.8, representing diffuse disease.

Exclusion Criteria:

1. Previously undergone percutaneous coronary intervention (PCI);
2. History of heart failure or myocardial infarction;
3. Acute myocardial infarction;
4. Primary or secondary cardiomyopathy;
5. Primary or secondary severe valvular heart disease;
6. Severe systemic infections;
7. Malignant cachectic diseases and an estimated survival of less than one year;
8. Patients who are currently participating in other clinical trials involving drugs or devices and have not yet reached the primary endpoint of those trials;
9. Patients whom the investigator deems to have other conditions that make them unsuitable for participation in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients with stable angina, unstable angina, suspected myocardial ischemia, or coronary artery stenosis of less than 50%, who do not have cardiomyopathy or obstructive epicardial coronary artery disease. Specifically, we will focus on two groups: (1) patients with caIMR values between 20 and 30, and (2) patients with diffuse disease.
Sampling Method: Non-Probability Sample
Enrollment: 508 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Patients' Seattle Angina Questionnaire (SAQ) scores | Before the procedure and six months post-procedure.
  The Seattle Angina Questionnaire (SAQ) is a rigorously validated disease-specific health status assessment tool widely used to evaluate symptoms, functional status, and quality of life in patients with coronary artery disease (CAD). Utilizing the SAQ as an endpoint in clinical trials ensures the scientific validity and comparability of study results, providing valuable insights for clinical practice.

SECONDARY OUTCOMES:
MACE (Major Adverse Cardiovascular Events) | At 6 months, 1 year, 2 years, and 3 years post-procedure.
  It is defined as a composite endpoint including cardiovascular death, target vessel revascularization, myocardial infarction, rehospitalization for angina, heart failure, and stroke.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608
- [Background] Chan PS, Jones PG, Arnold SA, Spertus JA. Development and validation of a short version of the Seattle angina questionnaire. Circ Cardiovasc Qual Outcomes. 2014 Sep;7(5):640-7. doi: 10.1161/CIRCOUTCOMES.114.000967. Epub 2014 Sep 2. PMID 25185249
- [Background] Kunadian V, Chieffo A, Camici PG, Berry C, Escaned J, Maas AHEM, Prescott E, Karam N, Appelman Y, Fraccaro C, Louise Buchanan G, Manzo-Silberman S, Al-Lamee R, Regar E, Lansky A, Abbott JD, Badimon L, Duncker DJ, Mehran R, Capodanno D, Baumbach A. An EAPCI Expert Consensus Document on Ischaemia with Non-Obstructive Coronary Arteries in Collaboration with European Society of Cardiology Working Group on Coronary Pathophysiology & Microcirculation Endorsed by Coronary Vasomotor Disorders International Study Group. Eur Heart J. 2020 Oct 1;41(37):3504-3520. doi: 10.1093/eurheartj/ehaa503. PMID 32626906
- [Background] Sara JD, Widmer RJ, Matsuzawa Y, Lennon RJ, Lerman LO, Lerman A. Prevalence of Coronary Microvascular Dysfunction Among Patients With Chest Pain and Nonobstructive Coronary Artery Disease. JACC Cardiovasc Interv. 2015 Sep;8(11):1445-1453. doi: 10.1016/j.jcin.2015.06.017. PMID 26404197
- [Background] Liu L, Abdu FA, Yin G, Xu B, Mohammed AQ, Xu S, Lv X, Luo Y, Zu L, Yang C, Zhang Z, Zhou Y, Cai H, Lv Z, Xu Y, Che W. Prognostic value of myocardial perfusion imaging with D-SPECT camera in patients with ischemia and no obstructive coronary artery disease (INOCA). J Nucl Cardiol. 2021 Dec;28(6):3025-3037. doi: 10.1007/s12350-020-02252-8. Epub 2020 Sep 30. PMID 33000403
- [Background] Radico F, Zimarino M, Fulgenzi F, Ricci F, Di Nicola M, Jespersen L, Chang SM, Humphries KH, Marzilli M, De Caterina R. Determinants of long-term clinical outcomes in patients with angina but without obstructive coronary artery disease: a systematic review and meta-analysis. Eur Heart J. 2018 Jun 14;39(23):2135-2146. doi: 10.1093/eurheartj/ehy185. PMID 29688324
- [Background] Zhang D, Lv S, Song X, Yuan F, Xu F, Zhang M, Yan S, Cao X. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention: a meta-analysis. Heart. 2015 Mar;101(6):455-62. doi: 10.1136/heartjnl-2014-306578. Epub 2015 Jan 30. PMID 25637372
- [Background] Huang D, Gong Y, Fan Y, Zheng B, Lu Z, Li J, Huo Y, Escaned J, Huo Y, Ge J. Coronary angiography-derived index for assessing microcirculatory resistance in patients with non-obstructed vessels: The FLASH IMR study. Am Heart J. 2023 Sep;263:56-63. doi: 10.1016/j.ahj.2023.03.016. Epub 2023 Apr 12. PMID 37054908
- [Background] Li J, Gong Y, Wang W, Yang Q, Liu B, Lu Y, Xu Y, Huo Y, Yi T, Liu J, Li Y, Xu S, Zhao L, Ali ZA, Huo Y. Accuracy of computational pressure-fluid dynamics applied to coronary angiography to derive fractional flow reserve: FLASH FFR. Cardiovasc Res. 2020 Jun 1;116(7):1349-1356. doi: 10.1093/cvr/cvz289. PMID 31693092